CLINICAL TRIAL: NCT06026449
Title: Effect of Gluten-free Diet on Clinical Symptoms, Immune Response and Microbiome in Primary Sclerosing Cholangitis and Inflammatory Bowel Disease
Brief Title: Gluten-free Diet in PSC and IBD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Jan Březina, Senior consultant, Institute for Clinical and Experimental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU22-06-00269
Record Dates: First submitted 2023-03-27; First posted 2023-09-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Sclerosing Cholangitis; Ulcerative Colitis; Biliary Tract Diseases; Biliary Disease Tract; Intestinal Disease
Keywords: Primary sclerosing cholangitis; Cholangitis; Gluten-free diet; Ulcerative Colitis; Microbiome
MeSH Terms: conditions — Cholangitis, Sclerosing; Colitis, Ulcerative; Biliary Tract Diseases; Intestinal Diseases; Cholangitis | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Prospective, self-controlled pilot clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary sclerosing cholangitis (Experimental)
  Interventions: Dietary Supplement: Gluten-free diet
- Ulcerative Colitis (Experimental)
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — After initial fase of habitual diet (6 months), patients will start Gluten-free diet for a period of 12 months

SUMMARY:
Primary sclerosing cholangitis (PSC) is a progressive disease of the biliary tree, which represents one of the most frequent indications for orthotopic liver transplantation (OLTx) in developed countries. There are several lines of evidence that dietary gluten/gliadin displays chronic pro-inflammatory, LPS-like properties. Recent evidence demonstrated the protective effect of gluten- free diet (GFD) in autoimmune diseases like type 1 diabetes, irritable bowel syndrome, non-celiac gluten sensitivity and some neurological disorders. This study is intended to explore therapeutic effect of GFD on PSC and IBD in prospective self-controlled mono-centric intervention study.

Hypothesis: Avoidance of gluten in diet will reduce progression, symptoms and intestinal inflammation in PSC and UC patients.

ELIGIBILITY:
Inclusion Criteria (for PSC group):

* Established diagnosis of PSC (based on radiologic features, typical finding on MRCP or ERCP)
* Age 18 - 65 years
* ALP 1,5x higher than ULN
* Signed informed consent

Exclusion Criteria (for PSC group):

* Patients on gluten-free diet
* Patients with coeliac disease or wheat allergy
* Liver transplant recipients
* PSC/AIH overlap syndrome
* Other causes of liver disease
* Radiologic or clinical signs of decompensated liver cirrhosis
* Advanced liver cirrhosis (MELD score ˃ 15)
* Recurrent acute cholangitis or cholangiogenic sepsis in past 3 months
* Use of antibiotics in past 3 months
* History of malignancy
* Pregnant women
* Not signed informed consent

Inclusion criteria (for UC group):

* Ulcerative colitis diagnosed based on clinical, endoscopic and histological findings
* Extension of affected colon > 15cm
* Mayo score 0-4
* Signed informed consent

Exclusion criteria (for UC group):

* CMV, Clostridium difficile enterocolitis in past 3 months
* Use of antibiotics in past 3 months
* Patients with coeliac disease or wheat allergy
* Patients on gluten-free diet
* Pregnant women
* Not signed informed consent
* Biologic therapy
* Methotrexate
* Prednison > 10 mg
* Not signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrease of laboratory markers of cholestasis | 6-12 months
  Change of alkaline phosphatase > 25% or normalisation.
Changes of intestinal microbiome composition. | 6-12 months
  16S-rRNA sequencing

SECONDARY OUTCOMES:
Changes of morphological signs of intestinal inflammation | 6-12 months
  Endoscopic Mayo score (Grade 0 - normal or inactive disease; Grade 1 - mild disease acitivity; Grade 2 - moderate disease acitivity; Grade 3 - Severe disease acitivity)
Improvement of quality of life and symptoms of ulcerative colitis. | 6-12 months
  UC Quality of life questionnaire (The Short Inflammatory Bowel Disease) Questionnaire)
Improvement of quality of life and symptoms of primary sclerosing cholangitis | 6-12 months
  PSC quality of life questionnaire (PSC PRO)
Changes of histopathological signs of intestinal inflammation | 6-12 months
  Nancy histological index (Grade 0 - no histological significant disease; Grade 1 - chronic inflammatory infiltrate with no acute inflammatory infiltrate; Grade 2 - Mildly active disease, Grade 3 - Moderately active disease; Grade 4 - Severly active disease)
Change from baseline of liver stiffness. | 6-12 months
  Shear-wave elastography (F0-F4)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of clinical and experimental medicine, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No